CLINICAL TRIAL: NCT04688047
Title: Urinary Incontinence and Transtheoretical Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevil Cicek Ozdemir, Research assistant, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KutahyaSCO
Record Dates: First submitted 2020-12-21; First posted 2020-12-29 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; transtheoretical model; motivational interviewing; nursing care
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Women aged 18 and over with urinary incontinence will be taken. A total of seven online interviews will be conducted with the women in the experimental group, one of which is pre-test, one is the last interview where the post-tests are applied, and five of which are motivational. Women in the experimental group were interviewed every 2 weeks and the women will be followed up by phone / mail every 2 weeks.
  Interventions: Behavioral: Nursing care based on the transtheoretical model
- Control (No Intervention): Women aged 18 and over with urinary incontinence will be taken. A total of two online interviews will be conducted with women in the control group, one of which is a pre-test interview and one is a final interview where post-tests are applied.

INTERVENTIONS:
Behavioral: Nursing care based on the transtheoretical model — Nursing care consists of urinary incontinence training, motivational interview and telephone/mail counseling processes.
  Arms: Experimental

SUMMARY:
The aim of the study is to evaluate the effectiveness of nursing care given online to women with urinary incontinence based on the Transtheoretical (Change) Model.

DETAILED DESCRIPTION:
The research was planned as a randomized experimental design with pre-test and post-test control groups. The research will be conducted in Kutahya, Turkey.

A total of seven online interviews will be conducted with the women in the experimental group, one of which is pre-test, one is the last interview where the post-tests are applied, and five of which are motivational. Women in the experimental group were interviewed every 2 weeks and the women will be followed up by phone/mail every 2 weeks. A total of two online interviews will be conducted with women in the control group, one of which is a pre-test interview and one is a final interview where post-tests are applied. No application will be made to women in the control group. All online calls to be made will be conducted via the WhatsApp application.

ELIGIBILITY:
Inclusion criteria

* 18 years or above
* Diagnosis of urinary incontinence according to the International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF)
* Mild to moderate incontinence according to the Incontinence Severity Index (ISI)
* Having a smartphone
* Using the WhatsApp application
* Being at one of the stages of pre-contemplation, contemplation, preparation, and action according to the evaluation form for stages of change
* Volunteering to participate in the study

Exclusion criteria

* Having risk factors that are thought to affect urinary incontinence (pregnancy; giving birth within the last year; having been diagnosed with recurrent urinary tract infection; having any health problem affecting the muscle and/or nervous system; having been diagnosed with a disease that increases intra-abdominal pressure and causes coughing, such as asthma, chronic obstructive pulmonary disease; using drugs that may cause urinary incontinence, such as diuretics, anticholinergics, antidepressants, antiparkinsonian, antihistamines, sedatives, narcotic analgesics for the past year; having been diagnosed with pelvic organ prolapse; receiving education and treatment for urinary incontinence in the last year)
* Being at the maintenance stage according to the evaluation form for stages of change
* Not volunteering to participate in the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
prevalence of urinary incontinence | Pre-interview (baseline) and last-interview 3 months after pre-interview (change from baseline at 3 months)
  Urinary incontinence according to International Consultation on Incontinence Questionnaire - Short Form
severity of urinary incontinence | Pre-interview (baseline) and last-interview 3 months after pre-interview (change from baseline at 3 months)
  Urinary incontinence severity according to Incontinence Severity Index

SECONDARY OUTCOMES:
Quality of life due to urinary incontinence | Pre-interview (baseline) and last-interview 3 months after pre-interview (change from baseline at 3 months)
  Quality of life due to urinary incontinence according to incontinence quality of life scale Incontinence quality of life scale scale consists of 22 questions in total. The questions are scored between 1 and 5 points. The minimum value that can be obtained from the scale is 22, the maximum value is 110. It is seen that the higher the score in this scale, the higher the quality of life of the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Senturk Erenel, Prof., Study Director — Gazi University
Locations (1):
- Kutahya Family Health Centers, Kütahya, Turkey (Türkiye)